CLINICAL TRIAL: NCT04265963
Title: CD123-Targeted CAR-T Cell Therapy for Relapsed/Refractory Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBC011
Record Dates: First submitted 2020-01-31; First posted 2020-02-12 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Leukemia; Leukemia, Myeloid; Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD123 CAR-T cells treat (Experimental): Patients will be be treated with CD123 CAR-T cells
  Interventions: Biological: CD123 CAR-T cells

INTERVENTIONS:
Biological: CD123 CAR-T cells — CD123 CAR-T cell therapy

SUMMARY:
There are limited options for treatment of relapse/refractory acute myeloid leukemia (AML). CD123 CAR-T cells may have an attractive and permanent effect on anti-tumor. This study purpose to estimate the safety and efficiency of CD123 CAR-T cells to patients with relapse/refractory AML.

DETAILED DESCRIPTION:
CD123 is expressed on most myeloid leukemia cells so it is a ideal target for CAR-T. Some researches have revealed that CD123 is a marker of leukemia stem cells, which indicates that the eradication of CD123 cells may prevent relapse of leukemia. In this study, investigators will evaluate the safety and efficacy of CAR-T targeting CD123 in patients with Acute Myelocytic Leukemia. The primary goal is safety and efficiency assessment, including adverse events and disease status after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent；
2. Diagnose as Relapsed/Refractory AML, and meet one of the following conditions：

   1. With persistent disease after at least two lines of therapy；
   2. Relapse to the last line of therapy in 6 months，as known as early recurrence;
   3. Relapse to the last line of therapy after 6 months, but refractory to this last line of therapy；
   4. Relapse more than once. The definition of relapse: Reappearance of blasts in the blood or bone marrow (>5%) or in any extramedullary site after a CR (the most common are CNS and testicular leukemia).
3. Evidence for cell membrane CD123 expression;
4. KPS>60;
5. The expect time of survive is above 3 months;
6. Ages: 2 to 75 years;
7. All genders;
8. The patients that diagnosis as high risks, relapse/refractory or inconformity criteria to other therapy；
9. No serious mental disorders;
10. Left ventricular ejection fraction ≥40%;
11. Sufficient hepatic function defined by ALT/AST<5 x ULN and bilirubin≤34.2μmol/L;
12. Sufficient renal function defined by creatinine clearance <220μmol/L;
13. Sufficient pulmonary function defined by indoor oxygen saturation≥92%;
14. No other illness may conflict with the protocol (e.g. autoimmune diseases, immune deficiency and organ transplantation；
15. Ability and willingness to adhere to the study visit schedule and all protocol requirements.

Exclusion Criteria:

1. Previous history of other malignancy;
2. Presence of uncontrolled active infection;
3. Evidence of disorder that need the treatment by glucocorticoids;
4. Active or chronic GVHD；
5. The patients treatment by inhibitor of T cell；
6. Pregnant or breasting-feeding women;
7. Any situation that investigators regard not suitable for attending in this study (e.g. HIV , HCVinfection or intravenous drug addiction) or may affect the data analysis.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events that related to treatment | 2 years
  Therapy-related adverse events will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0).
The response rate of CD123 CAR-T treatment in patients with relapse/refractory AML that treatment by CD123 CAR-T cells therapy | 2 years
  The response rate of CD123 CAR-T treatment will be recorded and assessed according to the National Comprehensive Cancer Network Guideline.

SECONDARY OUTCOMES:
Cellular kinetics of CD123 CAR-T in Blood | 2 years
  In vivo (peripheral blood) rate and quantity of CD123 CAR-T cells were determined by means of flow cytometry and qPCR
Cellular kinetics of CD123 CAR-T in Bone marrow | 2 years
  In vivo (bone marrow) rate and quantity of CD123 CAR-T cells were determined by means of flow cytometry and qPCR
Cellular kinetics of CD123 positive cells in Bone marrow | 1 years
  In vivo (bone marrow) rate and quantity of CD123 positive cells were determined by means of flow cytometry
Duration of Response (DOR) of CD123 CAR-T treatment in patients with refractory/relapsed AML | 2 years
  DOR will be assessed from the first assessment of CR or CRi to the first assessment of recurrence or progression of the disease or death from any cause (censored)
Progress-free survival(PFS) of CD123 CAR-T treatment in patients with refractory/relapsed AML | 2 years
  PFS will be assessed from the first CAR-T cell infusion to death from any cause or the first assessment of progression (censored)
Overall survival(OS) of CD123 CAR-T treatment in patients with refractory/relapsed AML | 2 years
  OS will be assessed from the first CAR-T cell infusion to death from any cause (censored)

CONTACTS AND LOCATIONS:
Overall Officials: Sanbin Wang, MD, Principal Investigator — 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China; Cheng Qian, PhD, Principal Investigator — Chongqing University Cancer Hospital
Locations (1):
- 920th Hospital of Joint Logistics Support Force, Kunming, Yunnan, China